CLINICAL TRIAL: NCT00877240
Title: The Influence of an Intervention Program on Altering Health Behavioral Patterns Among IDF's Staff
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of complaince
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Omer Ankol, MD, IDF's Medical Corps
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 735-2008
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Physical Fitness Habits; Balanced Nutrition; Weight Reduction; Smoking Cessation; Reduction of Stress
MeSH Terms: conditions — Weight Loss; Smoking Cessation

ARMS (1):
- Lifestyle counseling (Other)
  Interventions: Behavioral: Behavioral intervention-to determine the effectiveness of a general intervention on healthy living habits of IDF staff

INTERVENTIONS:
Behavioral: Behavioral intervention-to determine the effectiveness of a general intervention on healthy living habits of IDF staff — the program consists of 3 times a week of physical activity, nutrition advice, weight lodd program, stress workshop and smoking cessation workshop

SUMMARY:
The goal of this study is to determine the effectiveness of a general intervention that includes encouragement of physical activity and healthy living habits of officers and permanent staff in the IDF

ELIGIBILITY:
Inclusion Criteria:

* IDF'S staff member
* Age >26
* One or more risk factor

Exclusion Criteria:

* Cardio vascular condition
* Respiratory disease
* Other healthy conditions according to the physician's decision

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
physical fitness habits weight reduction balanced nutrition | one year

CONTACTS AND LOCATIONS:
Locations (1):
- IDF's Medical Corps, Tel Litwinsky, Israel